CLINICAL TRIAL: NCT02512276
Title: The Study of a Tele-pharmacy Intervention for Chronic Diseases to Improve Treatment Adherence (STIC2IT)
Brief Title: Tele-Pharmacy Intervention to Improve Treatment Adherence
Acronym: STIC2IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Vanguard Medical Associates (Other)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Niteesh K. Choudhry, MD, PhD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013P001076
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-03

CONDITIONS: Hyperlipidemia; Diabetes; Hypertension
Keywords: Medication Non-adherence; Hyperlipidemia; Diabetes; Hypertension
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus; Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telepharmacist intervention (Experimental): Patients diagnosed with diabetes, hypertension, or hyperlipidemia exhibiting sub-optimal adherence to their medications [defined as combined (average of averages) proportion of days covered (PDC) < 80%] who also have poor or worsening disease control.
  Interventions: Behavioral: Telepharmacist intervention
- Usual care (No Intervention): Patients randomized to this arm will receive usual care.

INTERVENTIONS:
Behavioral: Telepharmacist intervention — The intervention consists of a brief telephonic consultation with a clinical pharmacist using behavioral interviewing techniques tailored to patient's level of health activation and progress reports of medication-taking and disease control. Based on the barriers identified during the initial telephone consultation, patients will be offered more intensive support including reminder and motivational text-messages, video visits and pillboxes.
  Arms: Telepharmacist intervention

SUMMARY:
The purpose of this cluster randomized controlled trial is to evaluate whether a novel tele-pharmacist-based intervention for patients with hyperlipidemia, hypertension, and diabetes improves medication adherence, disease control, and patients' understanding of their treatment.

DETAILED DESCRIPTION:
Long-term adherence to evidence-based medications remains exceptionally poor. Half of all patients become non-adherent within a year of treatment initiation. Interventions that improve medication adherence may have important clinical benefits across large populations, and may even be cost-saving by reducing rates of costly and morbid clinical outcomes such as myocardial infarction and stroke.

The Study of a Tele-pharmacy Intervention for Chronic diseases to Improve Treatment adherence (STIC 2 IT) is a cluster randomized controlled trial (RCT) evaluating whether a novel tele-pharmacist-based intervention improves medication adherence and disease control among individuals with hyperlipidemia, hypertension, and diabetes who are nonadherent to their medications and who have poor or worsening disease control. The intervention consists of a brief telephonic consultation with a clinical pharmacist using behavioral interviewing techniques tailored to patient's level of health activation and progress reports of medication-taking and disease control. Based on the barriers identified during the consultation, patients will be offered more intensive support including reminder and motivational text-messages, video visits and pillboxes. Potentially eligible patients will be identified using data from paid-prescription claims data and the electronic health record. The study is being conducted at 14 practice sites in a large multi-specialty group practice with approximately 250 primary care physicians. Practice sites will be randomized to intervention or control. In intervention sites, the primary care physicians of potentially eligible patients will be asked whether they would like patients to be enrolled in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Filled and poorly adherent (defined as a PDC < 80%) to medication for hyperlipidemia, hypertension, or diabetes
* Suboptimal average adherence to all of the qualifying medications that a patient has filled (defined as combined (average of averages) PDC < 80%)
* For patients with hypertension or diabetes, poor or worsening disease control (according to relevant clinical targets)

Exclusion Criteria:

* Patients with <6 months of continuous enrolment in the health plan
* Patients with no available contact information

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4078 (Actual)
Dates: Start 2015-08; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Harvard Vanguard Medical Associates, Newton, Massachusetts, United States

REFERENCES:
- [Derived] Choudhry NK, Isaac T, Lauffenburger JC, Gopalakrishnan C, Lee M, Vachon A, Iliadis TL, Hollands W, Elman S, Kraft JM, Naseem S, Doheny S, Lee J, Barberio J, Patel L, Khan NF, Gagne JJ, Jackevicius CA, Fischer MA, Solomon DH, Sequist TD. Effect of a Remotely Delivered Tailored Multicomponent Approach to Enhance Medication Taking for Patients With Hyperlipidemia, Hypertension, and Diabetes: The STIC2IT Cluster Randomized Clinical Trial. JAMA Intern Med. 2018 Sep 1;178(9):1182-1189. doi: 10.1001/jamainternmed.2018.3189. PMID 30083727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telepharmacist Intervention | Usual Care
Started | 2038 | 2040
Completed | 2030 | 2029
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Population: Intention to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Telepharmacist Intervention | Usual Care | Total
Number analyzed (Participants) | 2038 | 2040 | 4078
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.7) | 59.2 (11.5) | 59.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 924 | 917 | 1841
  Male | 1114 | 1123 | 2237
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska | 4 | 2 | 6
  Asian | 94 | 95 | 189
  Black or African American | 579 | 448 | 1027
  Hispanic or Latino | 113 | 91 | 204
  Native Hawaiian or Other | 3 | 1 | 4
  Other | 68 | 95 | 163
  Patient Declined/ Missing | 84 | 72 | 156
  White | 1093 | 1236 | 2329
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2038 | 2040 | 4078

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: Average proportion of days covered (PDC) for medications to treat eligible conditions. An eligible condition is a diagnosis of either hyperlipidemia, hypertension, or diabetes and evidence of poor control for that condition at the time of enrollment. Adherence will be measured as an average of averages PDC only for medications that qualified a patient for inclusion in the study.
  Medication adherence is often reported as percentage of days covered.
Time Frame: 12 months
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: percentage of days covered
Arm/Group | Telepharmacist Intervention | Usual Care
Number analyzed (Participants) | 2038 | 2040
percentage of days covered | 46.2 (33.9) | 42.1 (33.8)
Statistical Analysis 1: Comparison: Telepharmacist Intervention vs Usual Care; Test type: Superiority; Mean Difference (Net) = 4.7, 95% CI 2-sided [3.0 to 6.4]

2. Secondary Outcome: Disease Control - All Eligible Conditions
Description: Percentage of patients achieving good disease control for all eligible conditions.
  Disease control was evaluated using laboratory or blood pressure values in the electronic health record and was based on clinical guideline targets (HbA1c values for patients with diabetes, systolic and diastolic blood pressure for patients with hypertension, and LDL values for patients with hyperlipidemia).
  This outcome measure disease control was measured as the proportion of patients achieving "good" disease control based on guideline-specified targets for all of their eligible conditions, as opposed to at least 1 for Outcome Measure 3. An eligible condition is a diagnosis of either hyperlipidemia, hypertension, or diabetes and evidence of poor control for that condition at the time of enrollment.
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Telepharmacist Intervention | Usual Care
Number analyzed (Participants) | 2038 | 2040
percentage of participants | 67.4 | 66.2
Statistical Analysis 1: Comparison: Telepharmacist Intervention vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.91 to 1.22]

3. Secondary Outcome: Disease Control
Description: Percentage of patients achieving good disease control for at least one eligible condition.
  Disease control was evaluated using laboratory or blood pressure values in the electronic health record and was based on clinical guideline targets (HbA1c values for patients with diabetes, systolic and diastolic blood pressure for patients with hypertension, and LDL values for patients with hyperlipidemia).
  This outcome measure disease control was measured as the proportion of patients achieving "good" disease control based on guideline-specified targets for all at least 1 eligible condition, as opposed to all of their eligible conditions for Outcome Measure 2. An eligible condition is a diagnosis of either hyperlipidemia, hypertension, or diabetes and evidence of poor control for that condition at the time of enrollment.
Time Frame: 12 months
Population: Intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | Telepharmacist Intervention | Usual Care
Number analyzed (Participants) | 2038 | 2040
percentage of participants | 72.9 | 71.2
Statistical Analysis 1: Comparison: Telepharmacist Intervention vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.10, 95% CI 2-sided [0.94 to 1.28]

4. Secondary Outcome: Healthcare Utilization - ER Visits
Description: Number of patients with at least 1 ER visit.
Time Frame: 12 months
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Telepharmacist Intervention | Usual Care
Number analyzed (Participants) | 2038 | 2040
Participants | 90 | 113
Statistical Analysis 1: Comparison: Telepharmacist Intervention vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.45 to 0.85]

5. Secondary Outcome: Healthcare Utilization - Office Visits
Description: Number of patients with at least 1 office visit.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telepharmacist Intervention | Usual Care
Number analyzed (Participants) | 2038 | 2040
Participants | 641 | 594
Statistical Analysis 1: Comparison: Telepharmacist Intervention vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.91 to 1.36]

6. Secondary Outcome: Healthcare Utilization - Hospitalizations
Description: Number of patients with at least 1 hospitalization.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Telepharmacist Intervention | Usual Care
Number analyzed (Participants) | 2038 | 2040
Participants | 170 | 156
Statistical Analysis 1: Comparison: Telepharmacist Intervention vs Usual Care; Test type: Superiority; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.78 to 1.34]

ADVERSE EVENTS:
Time Frame: We did not collect adverse event data (no investigational drug studied). Adverse events were not a pre-specified outcome for the trial. We also did not measure or evaluate mortality.
Description: We did not collect adverse event data (no investigational drug studied). Adverse events were not a pre-specific outcome for the trial. We also did not measure or evaluate mortality.
Arm/Group | Telepharmacist Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02512276/Prot_SAP_000.pdf